CLINICAL TRIAL: NCT05609877
Title: NON-pharmacological Approach Less Invasive Surfactant Administration (NONA-LISA) Trial: Protocol for a Randomised Controlled Trial
Brief Title: The NONA-LISA Trial
Acronym: NONA-LISA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Lise Aunsholt, MD, PhD, associate professor, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: The NONA-LISA trial
Record Dates: First submitted 2022-10-18; First posted 2022-11-08 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-07

CONDITIONS: Respiratory Distress Syndrome in Premature Infant
MeSH Terms: interventions — Sodium Chloride; Fentanyl

STUDY DESIGN:
Intervention Model Description: The randomisation will be stratified according to trial site and gestational age (GA) less than 28 or 28+ gestational weeks. Both groups will receive treatment by experienced teams of neonatal nurses and neonatologists. Both groups will receive the non-pharmacological approach as the basic treatment (part of routine).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participant, care provider, investigator and outcomes assessor will initially be blinded to treatment with analgesia or placebo (isotonic saline solution). Need for additional doses of analgesia will be decided according to section "Interventions" and will not be blinded. To reduce risk of interpretation bias, primary analyses will be performed blinded to the group allocation (Group A compared with Group B) and will be presented to all authors, who will agree on two alternative written interpretations before the randomisation code will be unblinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fentanyl group (Active Comparator): Patients will receive 0.5-1 mcg/kg fentanyl intravenously as pre-procedure analgesia for Less Invasive Surfactant Administration (LISA).
  The staff will perform LISA using standard pre- and post-procedure care, including non-pharmacological treatment and the use of atropine, caffeine, and naloxone at the clinician's discretion, based on local protocols and guidelines. All medications will be registered.
  Interventions: Procedure: Less Invasive Surfactant Administration (LISA); Drug: Fentanyl; Behavioral: Non-pharmacological standard operating procedure
- Saline group (Sham Comparator): Patients will receive a placebo (isotonic saline) instead of pre-procedure analgesia for Less Invasive Surfactant Administration (LISA).
  The staff will perform LISA using standard pre- and post-procedure care, including non-pharmacological treatment and the use of atropine, caffeine, and naloxone at the clinician's discretion, based on local protocols and guidelines. All medications will be registered.
  Interventions: Drug: Isotonic saline; Procedure: Less Invasive Surfactant Administration (LISA); Behavioral: Non-pharmacological standard operating procedure

INTERVENTIONS:
Drug: Isotonic saline — Isotonic saline will be administered intravenously instead of pre-procedure analgesia.
  Arms: Saline group
Procedure: Less Invasive Surfactant Administration (LISA) — All infants will be treated with the Less Invasive Surfactant Administration (LISA) procedure
Drug: Fentanyl — Fentanyl 0.5-1.0 mcg/kg will be administered intravenously as pre-procedure analgesia
  Arms: Fentanyl group
Behavioral: Non-pharmacological standard operating procedure — All infants will receive the same non-pharmacological standard operating procedure.

SUMMARY:
The NONA-LISA trial will be an investigator-initiated, multicentre, pragmatic, parallel-group, blinded RCT conducted at four university hospitals across Denmark. A total of 324 inborn premature infants will be included within 36 months at four neonatal intensive care units (NICUs) across Denmark (approximately 2 infants per month per unit).

The aim is to compare LISA using a non-pharmacological approach alone with routine analgesic treatment combined with a non-pharmacological approach (according to local guidelines) regarding LISA failure defined as the need for positive pressure ventilation for 30 min or more (cumulated) within 24 hours after the procedure in infants born prior to 30 gestational weeks.

DETAILED DESCRIPTION:
Background

Less Invasive Surfactant Administration (LISA) is a way of applying surfactant in the trachea by use of a catheter during spontaneous breathing and after applying nasal continuous positive airway pressure (nCPAP). However, use of pre-procedure analgesia with risk of apnoea may prevent LISA to achieve its full potential.

Aim

This study aims to compare the LISA procedure using a non-pharmacological approach to the LISA procedure using analgesic treatment with 0.5-1 mcg/kg fentanyl in infants born at 24 to 29 completed gestational weeks who fulfil the criteria for surfactant treatment.

Trial design

The NONA-LISA trial will be an investigator-initiated, multicentre, pragmatic, parallel-group, blinded RCT conducted at four university hospitals across Denmark. A total of 324 inborn premature infants will be included within 36 months at four neonatal intensive care units (NICUs) across Denmark (approximately 2 infants per month per unit).

Participants

Eligible infants will be born at 24+0 to 29+6 weeks of gestation at one of the trial sites meeting the criteria for first-choice surfactant treatment by LISA as described by Sweet et al.: worsening babies with RDS and FiO2 > 0.30 on CPAP pressure ≥6 cm H2O. Infants will be excluded if they have any of the exclusion criteria: 1) suspicion of lung hypoplasia, 2) endotracheal intubation at any time before randomisation, 3) suspicion of pneumothorax, pulmonary haemorrhage or pleural effusion before LISA, 4) major congenital anatomical anomalies as described by the European Surveillance of Congenital Anomalies (EUROCAT).

Interventions

The randomisation will be stratified according to trial site and gestational age (GA) less than 28 or 28+ gestational weeks. Both groups will receive treatment by experienced teams of neonatal nurses and neonatologists. Both groups will receive the non-pharmacological approach as the basic treatment (part of the routine). Additional analgesics will be provided at the clinician's discretion. Patients will receive the unit's standard pre-procedure and post-procedure care, and both procedures will use video laryngoscopes.

Participants in the control group will receive surfactant after receiving intravenous analgesics.

Participants in the intervention group (LISA using the non-pharmacological approach) will receive surfactant after receiving a similar volume of intravenous isotonic saline solution.

Outcomes

The primary outcome of this trial is the need for invasive ventilation, meaning mechanical or manual ventilation via an endotracheal tube for at least 30 min (cumulated) within 24 h of the procedure. Non-invasive ventilation (NIV) is not included in the primary outcome.

Sample size

We have calculated our sample size based on the primary outcome with an alpha of 5%, a power of 80%, and a ratio of 1:1 between intervention and control groups.

Based on previous studies, we anticipate an incidence of "positive pressure ventilation for at least 30 minutes (cumulated) within 24 hours after procedure" in the control group around 45%. Using 30% incidence reduction as anticipated intervention effect, we will need to randomise a total of 324 infants.

ELIGIBILITY:
Inclusion Criteria:

* Infants born at one of the trial sites with a gestational age of 24+0 to 29+6 weeks and meeting the criteria for first-choice surfactant treatment by LISA as described by Sweet et al.: worsening babies with RDS and FiO2 > 0.30 on CPAP pressure ≥6 cm H2O.

Exclusion Criteria:

1. suspicion of lung hypoplasia,
2. endotracheal intubation at any time before randomisation,
3. suspicion of pneumothorax, pulmonary haemorrhage or pleural effusion before LISA,
4. major congenital anatomical anomalies as described by the European Surveillance of Congenital Anomalies (EUROCAT).

Ages: 24 Weeks to 30 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 324 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
LISA failure within 24 hours. | 24 hours after procedure.
  The primary outcome will be LISA failure in terms of the need for endotracheal intubation and mechanical ventilation for at least 30 minutes (cumulated) within 24 hours after the procedure.

SECONDARY OUTCOMES:
Incidence of additional fentanyl administration | During the procedure, an average of 5-10 minutes.
  This will include the number of injection(s), dosage, cumulated dose, and indications defined as pain/discomfort/sedation/other.
Pain or discomfort during the procedure (according to COMFORTneo score >14). | 24 hours after procedure
  This will include a numerical and a categorical variable (COMFORTneo score >/< 14).
Bradycardia <100 BPM for a minimum duration of 4 seconds. | 24 hours after procedure.
  This is a categorical variable (yes/no).
Need for a second dose of surfactant | 24 hours after procedure.
  This is a categorical variable (yes/no).
Escalation from LISA to INSURE in the same attempt | 24 hours after procedure.
  This is a categorical variable (yes/no).
Apnoea that require bag and mask ventilation during the procedure | 24 hours after procedure.
  This is a categorical variable (yes/no).
Observed surfactant reflux | 24 hours after procedure.
  This is a categorical variable (yes/no).
Desaturation with SaO2 (right extremity measure) <85% during the procedure | 24 hours after procedure.
  This is a categorical variable (yes/no).
Procedural time consumption from the introduction of the laryngoscope blade into the oral cavity to removal of the catheter. | 24 hours after procedure.
  This is a categorical variable (yes/no).
Number of attempts of insertion of the catheter in the trachea. | 24 hours after procedure.
  This is a numerical variable.
Number of attempts of insertion of the laryngoscope in the oral cavity. | 24 hours after procedure.
  This is a numerical variable.
Time from meeting the criteria for surfactant treatment until surfactant administration | 24 hours after procedure.
  This is a numerical variable in minutes.
Incidence of endotracheal intubation. | 48 hours after procedure
  This is a categorical variable.
Incidence of pneumothorax within 48 hours after LISA. | 48 hours after procedure.
  This is a categorical variable.
Incidence of massive pulmonary haemorrhage within 48 hours after LISA (defined as the aspiration of haemorrhagic secretions from the trachea concurrent with the need for escalated respiratory support). | 48 hours after procedure.
  This is a categorical variable.
Incidence of in-hospital mortality before discharge. | Through study completion, an average of 6 months.
  This is a categorical variable.
Cumulated duration of mechanical ventilation during hospitalisation. | Before discharge (through study completion, an average of 6 months).
  This is a numerical variable.
Cumulated duration of positive pressure ventilation during hospitalisation. | Before discharge (through study completion, an average of 6 months).
  This is a numerical variable.
Incidence of escalation of respiratory support from CPAP to other NIV modes during hospitalisation. | Before discharge (through study completion, an average of 6 months).
  This is a categorical variable.
Cumulated duration of all types of non-invasive respiratory support during hospitalisation. | Before discharge (through study completion, an average of 6 months).
  This is a numerical variable.
Cumulated duration of oxygen treatment with fraction of inspired oxygen (FiO2) >0.21. | Before discharge (through study completion, an average of 6 months).
  This is a numerical variable.
Cumulated duration of any repisratory support during hospitalisation. | Before discharge (through study completion, an average of 6 months).
  This is a numerical variable.
Duration of hospitalisation. | Before discharge (through study completion, an average of 6 months).
  This is a numerical variable.
Incidence of necrotising enterocolitis (according to Bell's Staging Criteria). | Before discharge (through study completion, an average of 6 months).
  This is a categorical variable.
Incidence of treatment-demanding retinopathy of prematurity. | Before discharge (through study completion, an average of 6 months).
  This is a categorical variable.
Incidence of intraventricular haemorrhage grade 3-4 and periventricular leukomalacia. | Before discharge (through study completion, an average of 6 months).
  This is a categorical variable.
Composite outcome of death or moderate/severe BPD at 36 weeks of corrected gestational age. | 36 weeks of corrected gestational age.
  This is a categorical variable.

CONTACTS AND LOCATIONS:
Overall Officials: Niklas Breindahl, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (4):
- Denmark (4):
  - Neonatalafsnittet, Børn- og Ungeafdelingen, Reberbansgade 15, Aalborg
  - Department of Paediatrics (Intensive Care Neonatology) and Perinatal Research Unit, Aarhus
  - Department of Neonatal and Pediatric Intensive Care, Blegdamsvej 9, Copenhagen
  - H.C. Andersen Børne- og Ungehospital, Kløvervænget 23C, Indgang 60, Odense

IPD SHARING:
Plan to Share IPD: No
The datasets used and/or analysed during the current study will be available from the principal investigator on reasonable request after publication of results.

REFERENCES:
- [Background] Breindahl N, Henriksen TB, Heiring C, Bay ET, Haaber J, Salmonsen TG, Carlsen ELM, Zachariassen G, Agergaard P, Viuff AF, Bender L, Gronnebaek Tolsgaard M, Aunsholt L. NON-pharmacological Approach Less Invasive Surfactant Administration (NONA-LISA) trial: protocol for a randomised controlled trial. Pediatr Res. 2024 Sep;96(4):1084-1089. doi: 10.1038/s41390-023-02998-0. Epub 2024 Jan 11. PMID 38200325
- [Background] Breindahl N, Tolsgaard MG, Henriksen TB, Roehr CC, Szczapa T, Gagliardi L, Vento M, Stoen R, Bohlin K, van Kaam AH, Klotz D, Durrmeyer X, Han T, Katheria AC, Dargaville PA, Aunsholt L. Curriculum and assessment tool for less invasive surfactant administration: an international Delphi consensus study. Pediatr Res. 2023 Sep;94(3):1216-1224. doi: 10.1038/s41390-023-02621-2. Epub 2023 May 4. PMID 37142651
- [Derived] Breindahl N, Henriksen TB, Heiring C, Bay ET, Haaber J, Salmonsen TG, Agergaard P, Carlsen ELM, Tolsgaard MG, Aunsholt L. Can non-pharmacological comfort care replace fentanyl in LISA? The NONA-LISA feasibility study. Pediatr Res. 2025 Aug 2. doi: 10.1038/s41390-025-04310-8. Online ahead of print. PMID 40753114